CLINICAL TRIAL: NCT04801290
Title: Benefits and Limitations of Transjugular Intrahepatic Portosystemic Shunts (TIPS) in Patients With Decompensated Liver Cirrhosis
Brief Title: TIPS in Patients With Decompensated Liver Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: BM_84982019
Record Dates: First submitted 2021-02-26; First posted 2021-03-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Decompensated Liver Cirrhosis
Keywords: Portal hypertension; TIPS; Refractory ascites; Variceal bleeding; Liver cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Ascites; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TIPS insertion
  Interventions: Procedure: TIPS insertion

INTERVENTIONS:
Procedure: TIPS insertion — Patients are included in the registry if they receive a transjugular intrahepatic portosystemic shunt at Hannover Medical School and provide written informed consent.

SUMMARY:
This is a single center patient registry of patients receiving a transjugular intrahepatic portosystemic shunt (TIPS) at Hannover Medical School. By collecting and analyzing clinical data as well as blood samples, the overall aim is to optimize TIPS therapy (e.g. specify selection criteria).

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Indication for TIPS insertion
* Treatment at the Department of Gastroenterology, Hepatology and Endocrinology of Hannover Medical School
* Informed consent

Exclusion Criteria:

* Pregnancy or Lactation
* Age <18 years
* Lack of Informed consent
* Symptomatic anemia with Hb <7g/dl

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with decompensated liver cirrhosis and an indication for TIPS placement at Hannover Medical School.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
  Patients who die within 1 year
Occurrence of (Minimal) Hepatic Encephalopathy | 1 year
  Using the Portosystemic encephalopathy (PSE) syndrome test, critical flicker frequency (CFF) and animal naming test (S-ANT)
Change in Nutritional Status | 1 year
  Nutritional Status will be measured by hand grip strength (dynamometer) in kg
Change in Quality of Life | 1 year
  Using the questionnaire short-form 36 (SF36) (Score range 0-100, higher scores correspond to better quality of life)

SECONDARY OUTCOMES:
Change in inflammatory markers (e.g. cytokine) | 12 months
  Different cytokines and markers of bacterial translocation (e.g. LPS) are measured
Change in different metabolites using mass spectroscopy (metabolomics measurements) | 12 months
  More than 300 metabolites will be measured
Analysis of cellular immunity by collection of peripheral blood mononuclear cells (PBMCs) | 12 months
  Fluorescence activated cell sorting (FACS) analysis, genetics and in vitro stimulation assays will be performed
Analysis of stool samples | 12 months
  Analysis of the intestinal microbiome and metagenome analysis (shotgun sequencing)
Measurement of portal hypertension | 6 months
  Measurement of the hepatic venous pressure gradient (HVPG) to ensure the efficacy of the TIPS insertion

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maasoumy, PD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Sandmann L, Egge JFM, Tiede A, Ehrenbauer AF, Kabelitz MA, Rieland H, Mauz JB, Meyer BC, Wedemeyer H, Weissenborn K, Maasoumy B. Plasma Ammonia Levels Predict Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt Placement. United European Gastroenterol J. 2025 Sep;13(7):1171-1183. doi: 10.1002/ueg2.70095. Epub 2025 Aug 9. PMID 40782353
- [Derived] Kabelitz MA, Gairing SJ, Tiede A, Schleicher EM, Ahl LG, Wagner L, Zucker-Reimann F, Rieland H, Mauz JB, Weinmann-Menke J, Meyer BC, Pitton MB, Wedemeyer H, Galle PR, Sandmann L, Maasoumy B, Labenz C. Impact of Frailty on the Prognosis of Patients With Liver Cirrhosis Undergoing Insertion of a TIPS. Aliment Pharmacol Ther. 2026 Jan;63(1):109-118. doi: 10.1111/apt.70315. Epub 2025 Aug 1. PMID 40751304
- [Derived] Ehrenbauer AF, Schneider H, Stockhoff L, Tiede A, Lorenz C, Dirks M, Witt J, Gabriel MM, Wedemeyer H, Hinrichs JB, Weissenborn K, Maasoumy B. Predicting overt hepatic encephalopathy after TIPS: Value of three minimal hepatic encephalopathy tests. JHEP Rep. 2023 Jun 28;5(9):100829. doi: 10.1016/j.jhepr.2023.100829. eCollection 2023 Sep. PMID 37600959